CLINICAL TRIAL: NCT04224883
Title: Effect of Different Feeding Method on Gastrointestinal Function of Critical Patients
Acronym: DFM-GFC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Guang Yang, Director, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFM-GFC
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Gastrointestinal Dysfunction; Critical Illness; Nutrition Disorders
Keywords: gastrointestinal function; enteral feeding; critical
MeSH Terms: conditions — Critical Illness; Nutrition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 24-hours group (Active Comparator): The critical patients randomized to 24-hours group will be received enteral nutrition preparation by 24 hours of continuously pumping through stomach tube every day.
  Feeding will be started within 24 hours in admission of ICU. The time of therapy is 5 days.
  Interventions: Procedure: Continuously feeding
- 16-hours group (Experimental): The critical patients randomized to 16-hours group will be received enteral nutrition preparation by 16 hours of continuously pumping through stomach tube every day.
  Feeding will be started within 24 hours in admission of ICU. The time of therapy is 5 days.
  Interventions: Procedure: 16-hours feeding
- intermittent group (Experimental): The critical patients randomized to intermittent group will be received enteral nutrition preparations by four meals every day(08:00,12:00 18:00,22:00), each meal are pumped within 60min or 120min through stomach tube.Feeding will be started within 24 hours in admission of ICU. The time of therapy is 5 days
  Interventions: Procedure: intermittent feeding

INTERVENTIONS:
Procedure: Continuously feeding — Daily amount of feeding were continuously pumped for 24 hours. EN preparation pumping scheme was as follows: The initial pumping speed was average pumping volume of total enteral nutrition in one day, and gastric residual volumes is checked every 4 hours. If it is not tolerable, the speed of the pumping is reduced by half on the original speed. GRV<200mL were considered markers of good tolerance.Feeding intolerance was defined as GRV>200 mL. If GRV>500mL, EN was stopped and reassessed after 4 hours.
  Other Names: Continuously-feeding pumped in 24 hours
  Arms: 24-hours group
Procedure: 16-hours feeding — Daily amount of feeding were continuously pumped for 16 hours.EN preparation pumping scheme was as follows: The initial pumping speed was average pumping volume of total enteral nutrition in one day, and gastric residual volumes is checked every 4 hours.If it is not tolerable, the speed of the pumping is reduced by half on the original speed. GRV<200 mL were considered markers of good tolerance. Feeding intolerance was defined as GRV>200 mL. If GRV>500mL, EN was stopped and reassessed after 4 hours.
  Other Names: Continuously-feeding pumped in 16 hours
  Arms: 16-hours group
Procedure: intermittent feeding — Daily amount of feeding were divided into four meals, each meal are pumped within 60mins or 120mins through stomach tube. EN preparation pumping scheme was as follows: If the volume of each meal is less than or equal to 250ml(≤250ml), pump in within 60min, if volume is greater than 250ml(>250ml), pump in within 120min and gastric residual volumes is checked before each intermittent feeding. If it can be tolerated, the velocity of the pumping can be increased by half of the original speed.If it is not tolerable, the speed of the pumping is reduced by half on the original speed. GRV<200 mL were considered markers of good tolerance. Feeding intolerance was defined as GRV>200 mL. If GRV>500mL, EN was stopped and reassessed after 4 hours.
  Other Names: intermittent-feeding pumped
  Arms: intermittent group

SUMMARY:
The intestine is the most vulnerable target organ in septic patients and is the first to be damaged organ in multiple organ dysfunction syndrome(MODS).Therefore, improving intestinal motility and mucosal barrier function is critical to the treatment of sepsis. Many studies have shown that, early enteral nutrition(EN) in patients with sepsis helps prevent and treat intestinal dysfunction, reducing ICU mortality and length of stay in ICU. However, there is little research on feeding methods. In this study the investigators will compare the outcomes of different feeding methods: continuously-pumped in 24 hours, continuouslypumped in 16 hours and intermittently-pumped through the stomach tube. The aim of this study is to investigate the effects of different feeding methods on intestinal function in septic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Septic patients in Department of Critical Care Medicine, Guangdong Provincial Hospital of Chinese Medicine;
2. APACHE-Ⅱ score greater than 15 points;
3. Signing the informed consent.

Exclusion Criteria:

1. Fasting patients in the clinical, such as digestive tract perforation, bleeding or postoperative patients with gastrointestinal tract;
2. Allergic to enteral nutrition preparations;
3. Don't want to attend the test or not with the healer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The mean time(hours) that reach to the caloric goal in every group | First 5 days after intervention
  Caloric goals using 25 kcal/kg (ideal body weight) for caloric need calculated by a single nutritionist.

SECONDARY OUTCOMES:
The rate of onset of Gastric residual (%) | First 5 days after intervention
  The definition of gastric residual is that gastric residual volume more than 500 ml. Comparison of rate of gastric residual among three groups.
Abdominal pressure (mmHg) | baseline and 5th day
  Abdominal pressure measurement: through the bladder indirect pressure measurement method, first taking the supine position, emptying the bladder urine, secondly pouring 50ml saline into the balloon catheter, to the pubic symphysis as the base point, keeping the piezometric tube be perpendicular to the ground, then abdominal pressure can be obtained indirectly.
the rate of new onset pneumonia (%) | First 5 days after intervention
  Diagnosis of onset pneumonia is defined as two of the following clinical criteria were required. Fever (>38.3℃) or hypothermia (≤36.0℃), leukocytosis (>10×10E9 cells/liter) or leukopenia (≤4×10E9 cells/liter), purulent tracheal aspirate or sputum. The rate of onset pneumonia be counted in each group.
The rate(%) of people whom can reaching the caloric goal | First 5 days after intervention
  Caloric goals using 25 kcal/kg (ideal body weight) for caloric need calculated by a single nutritionist.

OTHER OUTCOMES:
length of ICU stay (in days) | up to 12 weeks
  length of ICU stay (in days)
ICU mortality rate (%) | 28 days after intervention
  ICU mortality rate (%)

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lagu T, Rothberg MB, Shieh MS, Pekow PS, Steingrub JS, Lindenauer PK. Hospitalizations, costs, and outcomes of severe sepsis in the United States 2003 to 2007. Crit Care Med. 2012 Mar;40(3):754-61. doi: 10.1097/CCM.0b013e318232db65. PMID 21963582
- [Result] Nieuwenhuijzen GA, Deitch EA, Goris RJ. The relationship between gut-derived bacteria and the development of the multiple organ dysfunction syndrome. J Anat. 1996 Dec;189 ( Pt 3)(Pt 3):537-48. PMID 8982828
- [Result] Pastores SM, Katz DP, Kvetan V. Splanchnic ischemia and gut mucosal injury in sepsis and the multiple organ dysfunction syndrome. Am J Gastroenterol. 1996 Sep;91(9):1697-710. PMID 8792684
- [Derived] Yang G, Deng A, Zheng B, Li J, Yu Y, Ouyang H, Huang X, Chen H. Effect of different feeding methods on gastrointestinal function in critical patients (DFM-GFC): study protocol for a randomized controlled trial. Trials. 2022 Oct 20;23(1):882. doi: 10.1186/s13063-022-06807-7. PMID 36266668